CLINICAL TRIAL: NCT03632174
Title: Clinical Study for the Evaluation and Comparison of Cutaneous Acceptability and the Efficacy of 2 Cosmetic Products, Under Normal Conditions of Use, in Adult Participants With Atopic Dermatitis
Brief Title: Evaluation and Comparison of 2 Cosmetic Investigational Products in Adults With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CSUB0167
Record Dates: First submitted 2018-08-01; First posted 2018-08-15 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Atopic Dermatitis
Keywords: Probiotic; Atopic Dermatitis; Lactobacillus reuteri
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Ointments

STUDY DESIGN:
Intervention Model Description: Comparison of two cosmetic products
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Ointment with L. reuteri (Experimental): Adult subjects presenting with mild-moderate Atopic Dermatitis
  Interventions: Other: Topical Ointment with L. reuteri
- Topical Ointment without L. reuteri (Experimental): Adult subjects presenting with mild-moderate Atopic Dermatitis
  Interventions: Other: Topical Ointment without L. reuteri

INTERVENTIONS:
Other: Topical Ointment with L. reuteri — Topical Ointment containing live Lactobacillus reuteri DSM17938 applied twice daily in dry areas of the entire body
  Other Names: Probiotic ointment A
  Arms: Topical Ointment with L. reuteri
Other: Topical Ointment without L. reuteri — Topical Ointment that does not contain Lactobacillus reuteri DSM17938 applied twice daily in dry areas of the entire body
  Other Names: Non Probiotic ointment B
  Arms: Topical Ointment without L. reuteri

SUMMARY:
The study consists in the application of 2 investigational products (one group per investigational product) under normal conditions of use, in adult participants with Atopic Dermatitis.

It is carried out on cosmetic products, with the aim to further confirm safety of these products

DETAILED DESCRIPTION:
Probiotics are live micro-organisms which when administered in adequate amounts can exert a health benefit on the host. This health-promoting effects of Lactobacillus reuteri have been extensively studied in the gastrointestinal tract but it is clear that other areas are also interesting for the use of probiotics.

Atopic Dermatitis is a relapsing inflammatory skin disease appearing on persons with a genetic predisposition of allergic pathology. AD generally starts in childhood, however in some cases can continue into adult hood, in at least 10% of cases. AD can effect a persons quality of life and in the chronic stage it can present with dry skin and lichenification.

Research has shown that probiotics have an antimicrobial, anti-inflammatory and barrier function effect, and could therefore be used on subjects with Atopic Dermatitis to relieve and protect.

ELIGIBILITY:
Inclusion Criteria:

* Participant has not been on a course of long term treatment in particular with aspirin, products containing aspirin, anti-inflammatories, antibiotics, antihistamines, corticoids
* Participant presenting with mild to moderate atopic dermatitis according to the definition of the UK Working Party's Diagnostic Criteria for Atopic Dermatitis (SCORAD index >25)
* Participant presenting with a current lesion of Atopic Dermatitis on defined area

Exclusion Criteria:

* Participant is pregnant, breast feeding or not willing to take the necessary precautions to avoid pregnancy during the study
* Participant having background of intolerance or allergy
* Participant not respecting the washout period during which a person may not be involved in any other biomedical research projects
* Participant having skin exposed to sunlight within 2 weeks preceding the inclusion
* Participant having modified his/her cosmetic habits during the last two weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Appraisal of Cutaneous acceptability of the investigational products by dermatologist investigator | 4 weeks
  Cutaneous acceptability is assessed on the basis of clinical examination of the skin for physical signs (erythema, oedema, dryness) linked to the use of the investigational product and also evaluation the functional signs (prickling, tightness, heating)

SECONDARY OUTCOMES:
Change in SCORAD index over 8 week period | baseline, at 4 and 8 weeks
  Clinical evaluation by the dermatologist investigator to assess change in skin conditions to each parameter of "SCORing Atopic Dermatitis" (SCORAD) (erythema, edema, xerosis) and participant symptoms: pruritus and sleep quality
Change in Local SCORAD index | baseline, at 4, and 8 weeks
  Change evaluated by the dermatologist investigator at each visit, on the recurrent lesion (defined area) and control area selected at baseline

OTHER OUTCOMES:
Appraisal of cosmetic acceptability of the investigational products by participant questionnaire | 4 weeks
  Cosmetic acceptability of the products through participant filling in questionnaire adapted to the products, elaborated in collaboration with the study monitor.
  The questionnaire will address functional and physical signs of a reaction (application frequency, nature, location, intensity, duration)
  Conclusion on cutaneous acceptability: Very good/ Good / Moderately Good / Bad

CONTACTS AND LOCATIONS:
Overall Officials: Burgert Jaques Van Wyk, MB, ChB, Principal Investigator — South African Medical Association
Locations (1):
- Unit 12B, Waverly Business Park, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenfeldt V, Benfeldt E, Nielsen SD, Michaelsen KF, Jeppesen DL, Valerius NH, Paerregaard A. Effect of probiotic Lactobacillus strains in children with atopic dermatitis. J Allergy Clin Immunol. 2003 Feb;111(2):389-95. doi: 10.1067/mai.2003.389. PMID 12589361